CLINICAL TRIAL: NCT05002309
Title: Treatment Interrupts Depression Early
Acronym: TIDE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIDE01
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: Severe mental illness
MeSH Terms: conditions — Depression; Mental Disorders | interventions — Cognitive Behavioral Therapy; Antidepressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychotherapy (Experimental): Cognitive-behavioural therapy
  Interventions: Behavioral: Cognitive-Behavioural Therapy
- Pharmacotherapy (Experimental): Antidepressant medication
  Interventions: Drug: Antidepressant medication

INTERVENTIONS:
Behavioral: Cognitive-Behavioural Therapy — 20 sessions of individual CBT are offered over 16 weeks, conducted 1-on-1, with a trained and supervised therapist. Participants will learn about the cognitive, behavioural, emotional, and environmental factors which contribute to maintaining their depression. They will apply skills to interrupt unhelpful cognitive and behavioural patterns and engage in guided exploration to improve self-understanding. CBT is a structured and collaborative treatment. Weekly "homework" will be used to maximize opportunities for practice and consolidation of new skills. The individual sessions can be combined with optional family/parent/partner sessions, depending on the situation and preferences of the participant. All sessions will be video-recorded to allow high-quality supervision, fidelity- and quality-assurance. This corresponds to evidence available for CBT for adolescents and young adults that is established as the best practice through rigorous trials.
  Other Names: CBT
  Arms: Psychotherapy
Drug: Antidepressant medication — The choice of antidepressants follows best-established evidence for treating depression in adolescents and young adults. We will offer treatment with fluoxetine, starting at 10mg a day, increasing to 20mg a day after 1 week if tolerated; a protocol established as safe and effective in adolescents and adults in multiple trials. Additional increases to 40 or 60mg will be possible based on positive effects and side-effects and clinical judgement, as recommended in this age group. In cases of intolerance or adverse reaction to fluoxetine, we will switch to sertraline (25-200mg) or escitalopram (5-20mg), two antidepressants licensed by the FDA for major depressive disorder in adolescents. Treatment will be optimized over 16 weeks, a time-frame comparable to the CBT arm. Pharmacotherapy will be managed and prescribed by qualified psychiatrists when starting treatment and reviewed after 1 week, 2 weeks and then in 2-weekly intervals for the remainder of the 16 weeks acute treatment period.
  Other Names: ADM
  Arms: Pharmacotherapy

SUMMARY:
The TIDE project aims to establish personal indicators for initial treatment choice for youth with first episode depression. Specifically, 100 adolescents and young adults (age 12 to 25) with untreated major depressive disorder of recent onset will be randomly allocated in 1:1 ratio to one of two evidence-based regimens for youth depression: (A) Individual cognitive-behavioural therapy; and (B) Optimized pharmacological treatment with an antidepressant. All participants will be offered active treatment for up to 1 year and follow-up for 2 years to establish short- and long-term outcomes, including change in depressive symptoms, maintenance of remission, core role functioning, achievement of educational, occupational and social milestones, and quality of life. Baseline characteristics including duration of untreated depression, pre-existing anxiety, attention-deficit/hyperactivity disorder, substance use, symptoms of reduced interest and activity, sleep, rhythm and melody of speech, brain function, history of childhood adversity, coping style, repetitive thinking, and family history of depression and bipolar disorder will be tested as potential moderators of outcome. Characteristics that differentially predict outcomes in those allocated to initial cognitive-behavioural therapy and those allocated to initial treatment with antidepressants will be combined into a personalized allocation algorithm.

DETAILED DESCRIPTION:
Design: TIDE is an open-label randomized trial with two parallel arms and long-term follow-up.

Participants: Youth and young adults with major depressive disorder will participate.

Recruitment: Young people aged 12 to 25 will be recruited through family physicians, child and adolescent mental health services (NSHA, IWK Central referral), student health, traditional advertisement (posters), and social media advertisement (Instagram, Facebook, Reddit, and Twitter).

Random allocation: Consenting eligible participants will be randomly allocated in 1:1 ratio to intervention A (cognitive-behavioral therapy) or intervention B (optimized antidepressant treatment), by an independent statistician using random blocks (block size 4 to 8), stratified by participant age (<18; ≥18). The allocation sequence will be held by a statistician at a separate location (the Research Methods Unit) and will remain concealed from the assessment and treatment team until the baseline assessment is completed.

Interventions: It is our aim to personalize the choice between established active treatments, not to test an active treatment against an inactive control. Therefore, the investigator will offer every participant entering the study an intervention that is established as safe and effective. Within the established interventions, the investigator chose two that have the largest amount of evidence for efficacy: cognitive-behavioural therapy and the antidepressant fluoxetine. These two interventions are at equipoise, meaning that the investigator has equally high expectation of treatment success from both approaches. Yet the two treatment strategies represent distinct choices, with intervention A relying on intensive psychological treatment and intervention B on optimized delivery of the best-established medication treatment for depression in youth.

Because the first episode of depression is a dynamic state with a variety of outcomes, the intervention will proceed in stages.

Stage 0: Lead in. Participants may enter the study at different stages of the first episode onset, with some starting at a point where the indications for treatment or eligibility criteria are uncertain or at a time when the participant is undecided on whether they need or want to start active treatment. To accommodate these early stages, there is a lead-in of 1-4 weeks to establish the diagnosis, assess severity and support the participant while deciding on whether they want to start active treatment. This stage will include up to four weekly meeting with a clinician (psychiatrist, psychologist, or CBT therapist) that may involve information gathering, information provision, risk monitoring and supportive contact, but no cognitive-behavioural therapy or pharmacotherapy. If the participant and the clinician agree that treatment is indicated, the participant can transition to Stage 1 (active intervention). Stage 0 is not randomized. If the participant recovers and no longer meets inclusion criteria or decides that they do not need active treatment, they may transition directly to Stage 3 (Follow-up).

Stage1: Active interventions. At this stage, all participants will be offered active treatment for depression. Radom allocation will occur at the beginning of Stage 1 and will determine whether the participant is offered Intervention A or Intervention B.

Intervention A: Cognitive-behavioural therapy (CBT). This intervention starts with a course of 20 sessions of individual CBT, offered over 16 weeks. The sessions will be conducted one-on-one, with a trained and supervised CBT therapist giving full attention to one participant at a time. Over the course of treatment participants will develop an understanding of the cognitive, behavioural, emotional, and environmental factors which contribute to maintaining their depression. They will learn and apply skills to interrupt unhelpful cognitive and behavioural patterns and engage in guided exploration to improve self-understanding. CBT is a structured and collaborative treatment and, as such, each session will follow a similar pattern and commence with a collaboratively set agenda. Weekly "homework" will be used to maximize opportunities for practice and consolidation of new skills with the aim of the participant being able to apply these skills well beyond the termination of therapy. The individual sessions can be combined with optional family/parent/partner sessions, depending on the situation and preferences of the participant. All sessions will be video-recorded to allow high-quality supervision, fidelity- and quality-assurance. This way of delivery corresponds to the best evidence available for CBT for adolescents and young adults that is established as the best practice through rigorous trials.

Intervention B: Antidepressant pharmacotherapy. The choice of antidepressants follows the best established evidence for treating depression in adolescents and young adults. The investigator will initially offer treatment with fluoxetine, starting at 10mg once daily and increasing to 20mg once daily after one week if tolerated, a protocol established as safe and effective in both adolescents and adults across multiple trials. Additional dose increases to 40 or 60mg will be possible based on balance of positive effects and side-effects and clinical judgement, consistent with recommendations in this age group. In cases of intolerance or adverse reaction to fluoxetine, the investigator will switch to sertraline (25 to 200mg) or escitalopram (5 to 20mg), the other two antidepressants licensed by the Food and Drug Administration for major depressive disorder in adolescents. The treatment with fluoxetine (or sertraline, or escitalopram) will be optimized over 16 weeks, a time-frame comparable to the CBT intervention. The investigator expects that most participants will only use the antidepressant for as long as required to minimized overall exposure to pharmacotherapy. Pharmacotherapy will be managed and prescribed by qualified psychiatrists, referred to as pharmacotherapists through this protocol. The pharmacotherapist will hold appointments when starting the treatment, after 1 week, two weeks and then in two-weekly intervals for the reminder of the 16 weeks acute treatment period.

Stage 2. Continuation treatment and cross-over options: After completion of a course of CBT or antidepressant, further decisions depend on the outcome of the initial treatment and will be personalized, based on a discussion between the participant and a clinician. If a full remission of depression is achieved, the next stage may involve continuation of the same treatment (up to 4 booster sessions of CBT, continued treatment with an antidepressant). If a remission is not achieved, the best recommended next step is the cross-over to (or the addition of) the other established treatment. Therefore, participants who received CBT in Stage 1 and did not reach remission will be offered treatment with an antidepressant, and participants who received the antidepressant in Stage 1 will be offered CBT. The decision of whether to continue Stage 1 treatment will be based on the balance of benefits and adverse effects for the participant. Participants who started antidepressant in Stage 1 and did not achieve full remission may decide to continue the antidepressant while also receiving CBT or to stop the antidepressant with coordinated support from the pharmacotherapist and the CBT therapist.

Stage 3: Follow-up. The investigators will follow participants once every 3 months for up to 2 years. The purpose of this follow-up stage is to monitor the stability of remission and functional outcomes. If the investigators identify re-emergence of depressive symptoms, the investigators will offer Stage 2 interventions or appropriate clinical referral as appropriate based on consultation with the principal investigator or other qualified psychiatrist. For participants who do not achieve remission in stages 1 and 2, the clinically advisable next steps may involve augmentation with additional treatment. Such augmentation treatment is beyond the scope of the present protocol. Participants will be allowed to remain in the follow-up stage even if they receive additional treatment through regular clinical services or additional studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-25 years
* Diagnosis of major depressive disorder, onset of the major depressive disorder within the last 12 months. Depression considered the most significant problem in need of treatment.
* An additional inclusion criterion for entering Stage 1 (active intervention) is a minimum moderate depression severity (CDRS-R≥40; MADRS≥20) that justifies the need for treatment. Individuals who fulfill general inclusion criteria but are below the depression severity threshold for active intervention will still be eligible to participate in follow-up assessments.
* Verbal ability sufficient to participate in psychological treatment.

Exclusion Criteria:

* Personal history of a manic or hypomanic episode, diagnosis of a psychotic disorder, pervasive developmental disorder or autism spectrum disorder, intellectual disability, mental disorders secondary to neurological or other medical condition, active substance use disorder.
* Previous trial of any treatment for major depressive disorder lasting 4 weeks or longer, current use of antipsychotic, antidepressant or mood-stabilizer medication.
* Recent (past 6 weeks) change in any psychotropic medication (including stimulants, hypnotics, anxiolytics) or receipt of 4 of more sessions of cognitive-behavioural therapy.
* Pregnancy or breastfeeding. If participants become pregnant or learn of pregnancies during the study, we will consult with Dr. Tanya Tulipan and jointly make the best decision for the participant with the option to either continue or end study treatment.
* No one will be excluded based on sex, gender, race, ethnicity, or living arrangements.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of depressive symptoms | 1-16 weeks
  The primary outcome measure at Stage 1 will be the severity of depressive symptoms, indexed with the Montgomery-Åsberg Depression Rating Scale (MADRS) total score. The MADRS is scored on a scale from 0-60, the higher the score the higher the severity of symptoms.
Severity of depressive symptoms | 16-32 weeks
  The primary outcome measure at Stage 2 will be the severity of depressive symptoms, indexed with the Montgomery-Åsberg Depression Rating Scale (MADRS) total score. The MADRS is scored on a scale from 0-60, the higher the score the higher the severity of symptoms.
Proportion of time spent depression free | 16-104 weeks
  At Stage 3 follow-up, the primary outcome will be the proportion of time spent depression free, defined as a score of 1 or 0 on Longitudinal Interval Follow-up Evaluation (LIFE).

SECONDARY OUTCOMES:
Self-reported measure of depression. | 1-104 weeks
  Secondary outcomes will include a self-reported measure of depression (Quick Inventory of Depressive Symptomatology: QIDS). The QIDS is scored on a scale from 0-27, the higher the score the higher the severity of depressive symptoms.
Self-reported measure of generalized anxiety. | 1-104 weeks
  Secondary outcomes will include a self-reported measures of anxiety (General Anxiety Disorder-7: GAD-7. The GAD-7 is scored on a scale from 0-21, the higher the score the higher the severity of symptoms.
Self-reported measure of social anxiety. | 1-104 weeks
  Secondary outcomes will include self-reported measures of social anxiety (Social Phobia Inventory: SPIN). The SPIN is scored on a scale from 0-68, the higher the score the greater the distress from symptoms.
Self-reported measures of general psychopathology. | 1-104 weeks
  Secondary outcomes will include self-reported measures of general psychopathology (Youth Experiences Tracker Instrument: YETI). The YETI is scored on a scale from 0-78, the higher the score the higher the severity of symptoms.
Self-reported measure of quality of life. | 1-104 weeks
  Secondary outcomes will include self-reported measure of quality of life (Quality of Life Enjoyment & Satisfaction Questionnaire: QLES-Q). The QLES-Q has a maximum score of 70, higher scores indicating greater life satisfaction and enjoyment.
Objective measures of psychopathology. | 1-104 weeks
  Objective measures of psychopathology (speech). A score from the acoustics and content of speech indicative of depressive symptomatology. Standard scale. Higher score indicates more severe symptoms.
Objective measure of physical activity. | 1-104 weeks
  Objective measure of physical activity with an actigraph. Single continuous score.Higher score indicates more activity, which is a positive outcome.
Objective measures of sleep. | 1-104 weeks
  Objective measure of total durarion of sleep with an actigraph.
Objective measures of educational progress. | 1-104 weeks
  Objective measures of educational progress using transcripts, grade completion, and graduation. A single score will be derived summarizing the educational progress relative to a normative sample of young people of similar age. Higher score indicates better educational achievement.

OTHER OUTCOMES:
Functioning score | 1-104 weeks
  Functioning will be defined as a continuous score on CCIS-R Columbia Child Impairment Scale - Revised (CCIS-R - 12-17 years) or Social and Occupational Functioning Assessment Scale (SOFAS - 18 years+), standardized for each age group. Higher score indicates better functioning.
Developmental milestones achievement | 1-104 weeks
  At stage 3, long-term functional outcomes will be the achievement of age-appropriate milestones defined as a number and timing of milestones achieved relative to the person's age and school grade.A single score will be derived summarizing the achievement of milestones relative to a normative sample of young people of similar age. Higher score indicates better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Uher, MD, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (2):
- Canada (2):
  - Nova Scotia Health, Halifax, Nova Scotia
  - Centre intégré universitaire de santé et de services sociaux de l'Ouest-de-l'Île-de-Montréal / Centre de Recherche Douglas (Montreal West Island IUHSSC / Douglas Research Center), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No